CLINICAL TRIAL: NCT00886353
Title: Double-blind, Placebo-controlled Dose-escalation Phase I Study With Recombinant Human Soluble Angiotensin Converting Enzyme 2 (rhACE2) APN01 in Healthy Volunteers
Brief Title: Safety and Tolerability Study of APN01 (Recombinant Human Angiotensin Converting Enzyme 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apeiron Biologics (Industry)
Responsible Party: Prof. Dr. Krähenbühl, Chefarzt klinische Pharmakologie & Toxikologie, Universitätsspital 4031 Basel
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APN01-1-01
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2009-12

CONDITIONS: Pulmonary Diseases; Cardiovascular Diseases; Kidney Diseases; Cancer Diseases
Keywords: RAS; ACE2; Cardiovascular; Pulmonary; Angiotensin II; Angiotensin 1-7
MeSH Terms: conditions — Lung Diseases; Cardiovascular Diseases; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APN01 (Active Comparator): Healthy volunteers will receive APN01
  Interventions: Biological: APN01
- Placebo (Placebo Comparator): Physiological saline administrated i.v.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: APN01 — APN01, a physiological formulation of recombinant human Angiotensin Converting Enzyme 2 administrated i.v.
  Arms: APN01
Other: Placebo — Physiological saline administrated i.v.
  Arms: Placebo

SUMMARY:
The purpose of this study is to define the dose for a Phase II study and to investigate safety and tolerability of intravenous administration of recombinant soluble human Angiotensin Converting Enzyme 2 in healthy volunteers.

DETAILED DESCRIPTION:
APN01-1-01 is a placebo controlled double blinded Phase I study composed of a single dose, dose escalation part followed by a multiple dosage part. The first four cohorts (four individuals each) will receive 100, 200, 400 and 800 µg/kg APN01 i.v. or placebo. Cohorts 5 and 6 (three individuals each) will receive three and six i.v. APN01 administrations daily, respectively. Planned dosage of the multiple dose part will be 400 µg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥18 years
* Use of acceptable form of birth control
* Willing to comply with study protocol
* No significant background illness
* Signed informed consent form

Exclusion Criteria:

* Significant hematological, renal, hepatic, metabolic, psychiatric or pulmonary diseases.
* Heart disease or elevated blood pressure.
* Any other significant disease that could interfere with the subject's ability to complete the protocol
* History of alcohol or drug abuse
* Abnormal urinalysis
* Pregnant or lactating female subjects
* Use of anticoagulants or antihypertensive drugs, particularly drugs interfering with the renin-angiotensin-aldosterone system, Obesity or anorexia (BMI <18 or >30)
* History of malignancy, except basal cell carcinoma of the skin, Known history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection or positive serology testing in the study screening procedures (except indicating immunization)
* Participation in a clinical trial within the last 30 days
* Any of the following laboratory abnormalities:

  * WBC 15% outside of normal limits
  * Hemoglobin 15% outside of normal limits
  * Platelets 15% outside of normal limits
  * Aspartate transferase (AST) or alanine transferase (ALT) above 15% outside of normal limits
  * Alkaline phosphatase above 15% outside of normal limits
  * Urea above 15% outside of normal limits
  * Creatinine above 15% outside of normal limits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability profile of APN01 when administered as a single dose / multiple dose i.v. in healthy volunteers. Measures: Blood chemistry, Hematology, Urinalysis, Adverse events, Vital signs including blood pressure, pulse, respiratory rate, ECG | 31 Days

SECONDARY OUTCOMES:
To obtain pharmacokinetic and pharmacodynamic data for APN01 and to investigate potential immunogenicity of APN01. Measures: Systemic rhACE2 concentration and activity, potential humoral immune response, Angiotensin II and Angiotensin 1-7 plasma levels. | 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Kraehenbuehl, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Haschke M, Schuster M, Poglitsch M, Loibner H, Salzberg M, Bruggisser M, Penninger J, Krahenbuhl S. Pharmacokinetics and pharmacodynamics of recombinant human angiotensin-converting enzyme 2 in healthy human subjects. Clin Pharmacokinet. 2013 Sep;52(9):783-92. doi: 10.1007/s40262-013-0072-7. PMID 23681967